CLINICAL TRIAL: NCT00915135
Title: A Double-Blind, Dose-Response, Cross-Over Study of TAK-375 With Chronic Insomnia (Phase II Study) -- Polysomnographic Evaluation
Brief Title: Efficacy and Safety of Ramelteon on Chronic Insomnia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: General Manager, Japan Development Center, Pharmaceutical Development Division
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-375-CCT-001; U1111-1115-2062 (Registry Identifier: WHO)
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2010-05

CONDITIONS: Chronic Insomnia
Keywords: Insomnia; Sleep Initiation and Maintenance Disorders; Drug Therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ramelteon QD and Placebo QD (25 possible combinations total) (Experimental)
  Interventions: Drug: Ramelteon and Placebo (25 possible combinations total)

INTERVENTIONS:
Drug: Ramelteon and Placebo (25 possible combinations total) — Randomized sequence over two consecutive nights for a total of five treatment periods to include the following:
  Ramelteon 4 mg, tablets, orally over two nights
  Ramelteon 8 mg, tablets, orally over two nights
  Ramelteon 16 mg, tablets, orally over two nights
  Ramelteon 32 mg, tablets, orally over two nights
  Ramelteon placebo-matching tablets, orally over two nights
  Other Names: Ramelteon; Rozerem; TAK-375

SUMMARY:
The purpose of this study is to determine the dose response of Ramelteon, once daily (QD), in Japanese subjects with Chronic Insomnia

DETAILED DESCRIPTION:
Complaints of sleep disorder are increasing with today's aging society and changing lifestyle. Sleep disorders not only impact one's activities of daily living, but also impede one's social life, leading to reduced productivity and sometimes accidents through carelessness.

Ramelteon is a melatonin-1 receptor agonist under global development by Takeda Chemical Industries, Ltd., Osaka, Japan, for the treatment of transient and chronic insomnia and for the treatment of Circadian Rhythm Sleep Disorders.

ELIGIBILITY:
Inclusion Criteria:

* Has primary chronic insomnia for at least 3 months.
* Has a mean latency of greater than or equal to 20 minutes on 2 consecutive polysomnography screening nights with no night less than 15 minutes, and has a mean of at least 60 minutes of wake time across 2 nights with no night less than 45 minutes.
* Has a habitual bedtime between 8:30 PM and 12:00 AM.
* Has a body mass index that is not less than 17, but less than 34.
* Females of childbearing potential who are sexually active must agree to use a medically accepted means of contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria:

* Has a history of psychiatric disorder (including depression and anxiety), seizures, drug addiction, sleep apnea, nocturnal myoclonus and/or mental retardation as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition.
* Has a history of alcohol abuse within the previous 2 years.
* Has a hepatic disease, and a significant neurological, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematological or metabolic disease.
* Has a known hypersensitivity to ramelteon or related compounds, including melatonin.
* Has a positive hepatitis panel including hepatitis A, hepatitis B or hepatitis C.
* Has any clinically abnormal findings as determined by a medical history, physical examination, electrocardiogram or clinical laboratory tests by the investigator or sub investigator.
* Has experienced 3 hours or more of jet lag within 7 days preceding the polysomnography screening.
* Has an apnea-hypopnea index (per hour of sleep) greater than or equal to 10 as seen on the first night of polysomnography screening.
* Has periodic limb movement with arousal index (per hour o sleep) greater than or equal to 10 as seen on the first night of polysomnography screening.
* Has participated in an excessive weight loss program that may have given influence on the evaluation of this study, or altered the participant's exercise routine within 30 days prior to double-blind study medication administration.
* Has had a clinically significant illness within 30 days prior to double-blind study medication administration.
* Has had sleep schedule changes required by employment (e.g., shift worker) within 3 months prior to double-blind study medication administration.
* The investigator or sub investigator judges the study subject inappropriate for participation because it is considered difficult to complete the study, or participating in the study will not be in the best interest of the subject.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2002-05; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Mean Latency to Persistent Sleep | Mean of Nights 1 and 2.

SECONDARY OUTCOMES:
Mean Total Sleep Time | Mean of Nights 1 and 2.
Sleep Efficiency | Mean of Nights 1 and 2
Awake Time after Persistent Sleep | Mean of Nights 1 and 2.
Percent of Total Sleep Time in NREM sleep Stage 1 | Mean of Nights 1 and 2.
Percent of Total Sleep Time in NREM sleep Stage 2 | Mean of Nights 1 and 2.
Percent of Total Sleep Time in NREM sleep Stage 3/4 | Mean of Nights 1 and 2.
Percent of Total Sleep Time in REM sleep Stage | Mean of Nights 1 and 2.
Latency to REM sleep stage | Mean of Nights 1 and 2.
Subjective Sleep Latency | Mean of Nights 1 and 2.
Subjective Total Sleep Time | Mean of Nights 1 and 2.
Subjective Sleep Quality | Mean of Nights 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

REFERENCES:
- See also: Rozerem Package Insert. — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI